CLINICAL TRIAL: NCT00025090
Title: Second UK Phase III Anal Cancer Trial: A Trial of Chemoradiation and Maintenance Therapy for Patients With Anal Cancer
Brief Title: Radiation Therapy Plus Fluorouracil With or Without Additional Chemotherapy in Treating Patients With Primary Anal Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University College London (UCL) Cancer Institute (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000068911; NCRI-ACT-II; EU-20056; UKCCCR-ACT-II; ISRCTN26715889
Record Dates: First submitted 2001-10-11; First posted 2003-01-27 (Estimated); Last update posted 2013-08-26 (Estimated); Status verified 2007-03

CONDITIONS: Anal Cancer
Keywords: stage I anal cancer; stage II anal cancer; stage IIIA anal cancer; stage IIIB anal cancer; squamous cell carcinoma of the anus; cloacogenic carcinoma of the anus; basaloid carcinoma of the anus
MeSH Terms: conditions — Anus Neoplasms; Anal Canal Carcinoma | interventions — Cisplatin; Fluorouracil; Mitomycin; Radiotherapy

INTERVENTIONS:
Drug: cisplatin
Drug: fluorouracil
Drug: mitomycin C
Radiation: radiation therapy

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to kill tumor cells. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining chemotherapy with radiation therapy may kill more tumor cells. It is not yet known if fluorouracil plus radiation therapy is more effective with or without additional chemotherapy in treating anal cancer.

PURPOSE: Randomized phase III trial to compare the effectiveness of fluorouracil plus radiation therapy with or without additional chemotherapy in treating patients who have primary anal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the response rates in patients with primary epidermoid anal cancer treated with radiotherapy and fluorouracil with either mitomycin or cisplatin and with or without maintenance therapy.
* Compare local control and prevention or delay of disease dissemination in patients treated with these regimens.

OUTLINE: This is randomized, open-label, multicenter study. Patients are randomized to one of four treatment arms.

All patients undergo radiotherapy daily 5 days a week for 5.5 weeks. All patients also receive fluorouracil IV continuously over days 1-4 and 29-32.

* Arm I: Patients receive mitomycin IV on day 1.
* Arm II: Patients receive cisplatin IV on days 1 and 29.
* Arm III: Patients receive mitomycin as in arm I and maintenance therapy comprising fluorouracil IV continuously over days 1-4 and cisplatin IV on day 1 beginning 4-8 weeks after completion of primary therapy and repeating once 3 weeks later.
* Arm IV: Patients receive cisplatin as in arm II and maintenance therapy as in arm III.

Patients are followed at 2 months, every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

Peer Reviewed and Funded or Endorsed by Cancer Research UK

PROJECTED ACCRUAL: A total of 600 patients (150 per treatment arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed primary epidermoid anal cancer

  * Squamous cell
  * Basaloid
  * Cloacogenic
* No adenocarcinoma, malignant melanoma, mucoepidermoid carcinoma, lymphoma, or microinvasive anal intraepithelial neoplasia (without evidence of invasive disease) in the anal canal or margin
* No metastatic disease

PATIENT CHARACTERISTICS:

Age:

* Not specified

Performance status:

* 0-2

Life expectancy:

* Not specified

Hematopoietic:

* WBC greater than 3,000/mm^3
* Platelet count greater than 100,000/mm^3
* Hemoglobin greater than 10 g/dL

Hepatic:

* Liver function tests no greater than 2 times normal

Renal:

* Glomerular filtration rate at least 50 mL/min

Cardiovascular:

* No cardiovascular disease
* No uncontrolled angina pectoris
* No heart failure
* No clinically significant cardiac arrhythmias

Other:

* HIV negative
* No other significant concurrent illness
* Not predominately bed-bound or frail
* No severe sepsis
* No other prior or concurrent cancer or illness that would preclude study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* Not specified

Endocrine therapy:

* Not specified

Radiotherapy:

* No prior radiotherapy to pelvis

Surgery:

* Not specified

Other:

* No prior therapy for anal cancer

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2001-03; Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Complete response rate at 6 months
Acute toxicity as measured up to 4 weeks after chemoradiation
Recurrence-free survival

SECONDARY OUTCOMES:
Colostomy rate
In field recurrence rate as measured by confirmed disease within radiation therapy field
Cause-specific and overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Roger D. James, MD, Study Chair — Maidstone Hospital
Locations (13):
- United Kingdom (13):
  - Northwick Park Hospital, Harrow, England
  - Ipswich Hospital, Ipswich, England
  - Cookridge Hospital, Leeds, England
  - Saint Bartholomew's Hospital, London, England
  - Cancer Research UK and University College London Cancer Trials Centre, London, England
  - James Cook University Hospital, Middlesbrough, England
  - Mount Vernon Cancer Centre at Mount Vernon Hospital, Northwood, England
  - Nottingham City Hospital, Nottingham, England
  - Royal Marsden - Surrey, Sutton, England
  - Southend University Hospital NHS Foundation Trust, Westcliff-on-Sea, England
  - Aberdeen Royal Infirmary, Aberdeen, Scotland
  - Velindre Cancer Center at Velindre Hospital, Cardiff, Wales
  - Cancer Research Centre at Weston Park Hospital, Sheffield